CLINICAL TRIAL: NCT01529710
Title: Safety and Efficacy of Mirazid for Schistosomiasis Treatment as Compared to Praziquantel: An Open-label Randomized Non-placebo-Controlled Study
Brief Title: Safety and Efficacy of Mirazid for Schistosomiasis Treatment
Acronym: PHAR0211
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharco Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mirazid2012
Record Dates: First submitted 2012-02-06; First posted 2012-02-09 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Schistosoma Hematobium Infection; Schistosomiasis Mansoni
Keywords: Schistosomiasis hematobium; Schistosomiasis mansoni
MeSH Terms: conditions — Schistosomiasis haematobia; Schistosomiasis mansoni | interventions — myrrh resin; Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirazid (Experimental): Mirazid is an antischistosomal drug available in the local Egyptian market since 2001 (Mirazid®). It originates from Myrrh a medicinal herb that has been used for thousands of years. Myrrh (Arabian or Somali Myrrh) is an oleo-gum resin, obtained from the stem of various species of Commiphora (Burseraceae) growing in northeast Africa and Arabia.
  Interventions: Drug: Myrrh
- Praziquantel (Active Comparator): Tablets
  Interventions: Drug: Myrrh

INTERVENTIONS:
Drug: Myrrh — Subjects will be treated by Mirazid as 600 mg oral (Soft Gelatin Capsules) for 6 consecutive days or 40mg/Kg body weight of Praziquantel as a single oral dose. Subjects will be evaluated for success of treatment at 12 weeks of treatment. Evaluation will be done by examining urine or stool samples for Schistosomiasis including egg counts for the positive cases.
  Other Names: Mirazid; Praziquantel; Shistosomiasis; Oral

SUMMARY:
Clinical Trial Phase:Phase III

Primary Objectives:

* Compare Mirazid and Praziquantel cure rates for both Schistosoma species.
* Compare Mirazid and Praziquantel effect in lowering the intensity of infection for both Schistosoma species.

Secondary Objective:Identify and compare the types and severity of side and adverse effects between the Mirazid and Praziquantel.

Study Population:200 Schistosomiasis infected persons of both types of Schistosomiasis aged from 15-35 years. Those subjects will be selected from among those screened.Subjects will include both genders excluding chronically ill such as chronic liver disease patients and those with both types of Schistosomiasis.

Recruitment Period:3 months and subjects follow up for another 3 months followed by 3 months for statistical analysis and report writing Study Duration: Total study duration is expected to be 9 months: 3 months for recruitment, 3 months for follow up and 3 months for data management and report writing.

Endpoints: Will be measured at 3 months of successful administration of treatment either Mirazid or Praziquantel as per the randomization scheme. By then, final assessment of the response to treatment will be done by examining urine or stool of the subject for presence of Schistosoma eggs and its density if found.

Three negative urine or stool samples collected 2-days apart at 12 weeks post treatment will indicate treatment success. One positive sample collected at week 12 will indicate infection with Schistosomiasis.

DETAILED DESCRIPTION:
Study Design:This is a phase III, open-label randomized non-placebo-controlled Study in which the investigators will compare the efficacy and safety of Mirazid to Praziquantel as a treatment for Schistosomiasis. After screening, positive subjects for one of the Schistosomiasis will be recruited in the study. They will be treated by Mirazid as 600 mg oral (Soft Gelatin Capsules) for 6 consecutive days or 40mg/Kg body weight of Praziquantel as a single oral dose. Subjects will be evaluated for success of treatment at 12 weeks of treatment. Evaluation will be done by examining urine or stool samples for Schistosomiasis including egg counts for the positive cases.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent and young adults aged 15-30 years
* Positive for Schistosoma infection of any type.

Exclusion Criteria:

* Mixed Schistosoma infection of both types
* History of administration of treatment for Schistosoma infection in the last 6 months prior to the study.
* Severely ill patients
* Advanced chronic liver disease.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Compare Mirazid and Praziquantel cure rates for both Schistosoma species, and effect in lowering the intensity of infection for both Schistosoma species. | 9 months

SECONDARY OUTCOMES:
Identify and compare the types and severity of side and adverse effects between the Mirazid and Praziquantel. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ayat A Haggag, MD, Principal Investigator — Ministry of Health
Locations (2):
- Egypt (2):
  - Tanta Health Unit, Gharbiya
  - Health Unit of Atfeeh, Giza